CLINICAL TRIAL: NCT01068626
Title: A 26-week, Single Center, Randomized, Placebo-controlled, Double-blind, Parallel-group Study to Evaluate the Effect of Rosuvastatin on Visceral Adipose Tissue in Male Patients With Abdominal Obesity
Brief Title: Rosuvastatin in Visceral Adiposity
Acronym: RIVIERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 990312
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2011-03-02 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Placebo for Rosuvastatin (Placebo Comparator)
  Interventions: Drug: Placebo for rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg once daily
  Other Names: Crestor®
  Arms: Rosuvastatin
Drug: Placebo for rosuvastatin — once daily
  Arms: Placebo for Rosuvastatin

SUMMARY:
The purpose of this study is to investigate whether 6 months treatment with the cholesterol-lowering drug rosuvastatin may reduce visceral fat tissue in obese middle aged men.

DETAILED DESCRIPTION:
The accumulation of intra-abdominal fat has been suggested to be of primary importance in the development of the metabolic syndrome and associated metabolic disturbances and it has been hypothesized that a selective reduction of visceral fat tissue would improve the symptoms of the metabolic syndrome. Treatment with statins decrease levels of LDL-cholesterol and reduce coronary artery disease (CAD) events. Although it is widely accepted that the majority of benefit obtained with statins is a direct result of their lipid-lowering properties, they also demonstrate additional cholesterol-independent or pleiotropic effects. The results of experimental studies have now shown that statins decrease fat mass in the visceral region in an animal model. In the present study, we will investigate whether statins can decrease visceral obesity in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 40 and 65 years of age.
* Abdominal obesity
* Dyslipidemia
* Written informed consent.

Exclusion Criteria:

* Uncontrolled hypertension
* Diabetes mellitus
* Severe liver disease
* Severely reduced renal function
* Uncontrolled endocrine disorders
* History of or ongoing malignant disease
* Patients with known myopathic disease
* Recent alcohol or drug abuse
* Weight loss or weight gain during the three months prior to screening.
* Ongoing treatment with statins
* Ongoing treatment with calcineurin-inhibitors
* Ongoing treatment with anti-inflammatory drugs
* Received an investigational drug within 30 days prior to screening.
* Strong clinical indication for statin treatment
* In the Principal Investigator's opinion, the patient has other clinically significant cardiac, oncologic, neurologic or psychiatric disease that could be adversely affected by Study participation.
* For any reason the patient is considered by the Principal Investigator to be an unsuitable candidate to participate in the Study.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John-Olov Jansson, Prof, Study Chair — Department of Endocrinology, University of Gothenburg; Claes Ohlsson, Professor, Study Chair — Department of Clinical Pharmocology, University of Gothenburg; Anna Nilsson, MD, PhD, Study Chair — Department of Endocrinology, University of Gothenburg; Kristjan Karason, MD, PhD, Principal Investigator — Department of Molecular and Clinical Medicine at University of Gothenburg
Locations (1):
- Department of Molecular and Clinical Medicine, Sahlgrenska Academy at University of Gothernburg, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2006 to July 2007 a total of 78 subjects were screened at the Sahlgrenska Hospital. Among these, 59 fulfilled all inclusion and no exclusion criteria and were randomized to treatment. During follow-up 5 patients (7 %) withdrew from the study, resulting in 54 patients who completed the study, comprising 27 patients in each study group.
Pre-assignment Details: Among patients that were screened 19 patients did not fulfill inclusion criteria or displayed exclusion criteria and did not enter the study.
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Started | 30 | 29
Completed | 27 | 27
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (5.2) | 55 (4.1) | 54 (4.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 30 | 29 | 59
Region of Enrollment [Number; unit: participants]
  Sweden | 30 | 29 | 59
Weight [Mean (Standard Deviation); unit: kg] | 100 (12) | 100 (13) | 100 (13)
Height [Mean (Standard Deviation); unit: m] | 1.82 (0.06) | 1.80 (0.07) | 1.81 (0.07)
Hypertension [Number; unit: participants]
  YES | 8 | 7 | 15
  NO | 22 | 22 | 44
Current smoker [Number; unit: participants]
  YES | 3 | 6 | 9
  NO | 27 | 23 | 50
Visceral adipose tissue area [Mean (Standard Deviation); unit: cm2] — Visceral adipose tissue area measured with CT at the level of the fourth lumbar vertebrae.
  cm2 | 221 (66) | 219 (73) | 220 (69)
Subcutaneous adipose tissue area [Mean (Standard Deviation); unit: cm2] — Subcutaneous adipose tissue area measured with CT at the level of the fourth lumbar vertebrae.
  cm2 | 289 (69) | 310 (101) | 300 (86)
Visceral/subcutaneous adipose tissue area ratio [Mean (Standard Deviation); unit: ratio] | 0.79 (0.25) | 0.75 (0.27) | 0.77 (0.26)
Liver density [Mean (Standard Deviation); unit: Hounsfield units] — Liver density measured by computed tomography
  Hounsfield units | 52 (10) | 49 (14) | 50 (12)
LDL cholesterol [Mean (Standard Deviation); unit: mmol/L] | 3.59 (0.78) | 3.77 (0.79) | 3.69 (0.74)
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] | 5.3 (0.5) | 5.3 (0.5) | 5.3 (0.5)
Fasting insulin [Mean (Standard Deviation); unit: IU] | 12 (4.8) | 13 (9.4) | 12 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visceral Adipose Tissue Area Measured by Computed Tomography.
Time Frame: 6 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
cm2 | -1.5 (27) | 2.8 (26)

2. Secondary Outcome: Change in Subcutaneous Adipose Tissue Area
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
cm2 | 10 (34) | 1 (15)

3. Secondary Outcome: Change in the Ratio Between Intra-abdominal and Subcutaneous Tissue Area Measured by CT.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
ratio | -0.02 (0.11) | 0.01 (0.08)

4. Secondary Outcome: Change in Hepatic Fat Infiltration Measured by CT.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
Hounsfield units | 0 (5.2) | -2 (5.0)

5. Secondary Outcome: Change in Body Weight
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
kg | 0.2 (2.6) | 0.5 (1.5)

6. Secondary Outcome: Change in LDL
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Number analyzed (Participants) | 27 | 27
mmol/L | -1.4 (0.9) | -0.1 (0.9)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin | Placebo for Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 3/30 | 1/29
Other Adverse Events (participants affected / at risk) | 3/30 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=30) | Placebo for Rosuvastatin (N=29)
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=30) | Placebo for Rosuvastatin (N=29)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications during 3 months prior to public release and can embargo communications regarding trial results for an additional period of 3 months from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo